CLINICAL TRIAL: NCT06122597
Title: A Clinical Trial to Evaluate the Efficacy of ConcenTrace to Buffer pH Levels Within the Body.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trace Minerals (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20352
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: pH

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test arm: ConcenTrace (Experimental): Participants should follow this weekly dosing schedule:
  Week 1 - Days 1-3: take 5 drops of ConcenTrace with 8 oz of water or flavored water. Days 4-7: take 5 drops of ConcenTrace 2x daily with 8 oz of water or flavored water.
  Week 2: Take 10 drops of ConcenTrace 2x daily with 8 oz of water or flavored water.
  Week 3: Take 15 drops of ConcenTrace 2x daily with 8 oz of water or flavored water.
  Weeks 4-12: Take 20 drops of ConcenTrace 2x daily with 8 oz of water or flavored water.
  Interventions: Other: ConcenTrace

INTERVENTIONS:
Other: ConcenTrace — The product contains concentrated seawater from Utah's inland sea.

SUMMARY:
This virtual single-arm trial will last 12 weeks. Participants will take the drops daily and complete questionnaires at Baseline, Week 4, Week 8, and Week 12.

Urine pH measurements will be taken at Baseline, Week 4, Week 8, and Week 12 using pH test strips.

ELIGIBILITY:
Inclusion Criteria:

* Male or female. Aged 18+. Generally healthy - don't live with any uncontrolled disease. Willing to maintain their standard dietary pattern, activity level, and body weight for the duration of the study.

Exclusion Criteria:

* Anyone with a pre-existing chronic condition that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.

Anyone with known severe allergic reactions. Women who are pregnant, breastfeeding, or attempting to become pregnant. Anyone unwilling to follow the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in urine pH levels. [Timeframe: Baseline to Week 12] | 12 weeks
  Participants will use pH test strips to measure urine pH. Changes in urine pH will be evaluated.

SECONDARY OUTCOMES:
Change in score on the Metabolic Screening Questionnaire. | 12 weeks
  A Metabolic Screening Questionnaire (MSQ) was developed by the Toronto Centre for Naturopathic Medicine. The symptoms represented on a MSQ represent symptoms commonly associated with inflammation and toxicity. Participants will rate frequency and intensity of applicable symptoms according to the following scores:
  * Absent or rare symptoms - 0 points
  * Occasional, mild symptoms - 1 point
  * Occasional, severe symptoms - 2 points
  * Frequent, mild symptoms - 3 points
  * Frequent, severe symptoms - 4 points

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States